CLINICAL TRIAL: NCT03994302
Title: Monitoring the Antiphospholipid Syndrome:TOXicity of Drugs (APSTOX)
Acronym: APSTOX
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-19-10
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Antiphospholipid Syndrome; Immune Disease; Adverse Drug Event; Drug Toxicity
MeSH Terms: conditions — Antiphospholipid Syndrome; Immune System Diseases; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Immune toxicity induced by drugs and chemotherapies: Immune toxicity induced by drugs and chemotherapies Case reported in the World Health Organization (WHO) of immune toxicities(such as Antiphospholipid syndrome) of patient treated by a drug, with a chronology compatible with the drug toxicity
  Interventions: Drug: Drug inducing antiphospholipid syndrome

INTERVENTIONS:
Drug: Drug inducing antiphospholipid syndrome — Drugs susceptible to induce immune toxicities such as antiphospholipid syndrome

SUMMARY:
Several drugs and chemotherapies seem to have an impact on the immune system. This study investigates reports of immune toxicities such as antiphospholipid syndrome, including the International classification of disease ICD-10 for treatments in the World Health Organization (WHO) global Individual Case Safety Report (ICSR) database (VigiBase).

DETAILED DESCRIPTION:
Several drugs and chemotherapies seem to have an impact on the immune system and are responsible of a wide range of immune side effects such as antiphospholipid syndrome. Those are poorly described, due to the modificationof the pharmacopeia, and the recent recognition of several of these adverseevents.

This study investigates the main characteristics of patients affected by immune side effects imputed to drugs in particular antiphospholipid syndrome.

A causality assessment according to the WHO-UMC (World Health Organization - Uppsala Monitoring Center) is systematically applied.

ELIGIBILITY:
Inclusion Criteria:

- Case reported in the WHO's pharmacovigilance database till 01/06/2019

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with a drug that could be reported in the WHO's pharmacovigilance database
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
Immune toxicities (such as Antiphospholipid Syndrome) of drugs Identification and report of immune toxicities associated with drugs. | 01/06/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports

SECONDARY OUTCOMES:
Causality assessment of reported metabolic toxicities events according to the WHO system Case reported in the World Health Organization (WHO) database of individual safety case reports | 01/06/2019
Description of the type of immune toxicity depending on the category of drug Case reported in the World Health Organization (WHO) database of individual safety case reports | 01/06/2019
Description of the other immune related adverse events concomitant to the immune toxicity induced by drugs Case reported in the World Health Organization (WHO) database of individual safety case reports | 01/06/2019
Description of the duration of treatment when the toxicity happens (role of cumulative dose) Case reported in the World Health Organization (WHO) database of individual safety case reports | 01/06/2019
Description of the drug-drug interactions associated with adverse events Case reported in the World Health Organization (WHO) database of individual safety case reports | 01/06/2019
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed Case reported in the World Health Organization (WHO) database of individual safety case reports | 01/06/2019
Description of the population of patients having hematological toxicity adverse event Case reported in the World Health Organization (WHO) database of individual safety case reports | 01/06/2019

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gerardin C, Bihan K, Salem JE, Khachatryan H, Gerotziafas G, Fain O, Mekinian A. Drug-induced antiphospholipid syndrome: Analysis of the WHO international database. Autoimmun Rev. 2022 May;21(5):103060. doi: 10.1016/j.autrev.2022.103060. Epub 2022 Feb 1. PMID 35114404